CLINICAL TRIAL: NCT03390309
Title: Evaluation of A Partially Hydrolyzed Whey Protein Infant Formula in Improving Functional Gastrointestinal Disorders (FGIDs) Symptoms
Brief Title: Evaluation of A Partially Hydrolyzed in Improving FGIDs Symptoms
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Fudan-AN 001
Record Dates: First submitted 2017-11-26; First posted 2018-01-04 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-07

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Partially Hydrolyzed Formula (Other): Infant was identified and got 1 or more scores by using infant feeding & stool pattern questionnaire at Visit 1 will be assigned into experimental group randomly
  Interventions: Other: Partially Hydrolyzed Formula
- Normal Formula (Placebo Comparator): Normal Formula
  Interventions: Other: Normal Formula

INTERVENTIONS:
Other: Partially Hydrolyzed Formula — Partially Hydrolyzed Whey Protein Infant Formula
  Arms: Partially Hydrolyzed Formula
Other: Normal Formula — Normal Formula
  Arms: Normal Formula

SUMMARY:
Evaluation of A Partially Hydrolyzed Whey Protein Infant Formula in Improving Functional Gastrointestinal Disorders (FGIDs) Symptoms

DETAILED DESCRIPTION:
This study will investigate the prevalence of Shanghai area's infant with FGIDs symptom and contrast for the FGIDs symptoms by using different intervention means, and evaluate the effectiveness of FGIDs symptoms in infants by using partially hydrolyzed whey protein and low lactose infant formulation.

ELIGIBILITY:
Inclusion Criteria:

* Infants is formula-fed or mixed feeding a cow milk protein-based formula for less 7 days prior to enrollment.
* Infant is between 30-180 days of age.
* Infant's parent(s) or Legally authorized representative(LAR) has voluntarily signed and dated an informed consent form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) prior to any participation in the study.

Exclusion Criteria:

* Complementary food was added for infants or parents are willing to add complementary food during study.
* Suffer from infection/illness.
* Infant has suspected or known metabolic or physical diseases affecting infant feeding and/or metabolism.
* Infant has visible bloody stools (detected before enrollment) prior to enrollment.
* Participation in another study.

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-07-05 (Estimated); Primary Completion 2018-12-30 (Estimated); Study Completion 2019-06-28 (Estimated)

PRIMARY OUTCOMES:
Change of total symptom score of infant feeding & stool pattern questionnaire. | From enrollment to end of treatment（1 week）. The scores will be measured at the following time point: enrollment,end of treatment(one week after the start of treatment).
  Investigator report questionnaire. Total score consists of 6 sub scores based on different symptom scaleing : diarrhea(0= no; 1= yes), constipation(0= no; 1= yes), galactorrhea/spit milk(0= no; 1= yes), Irritability or crying(0= no; 0.5= yes), bloating/ tummy drum/ exhaust(0= no; 1= yes), other(0= no, 0.5=yes).